CLINICAL TRIAL: NCT04630145
Title: A Phase 2/3, Multicenter, Randomized, Open-label, Active-controlled Study to Evaluate the Efficacy and Safety of Bedaquiline Administered as Part of a Treatment Regimen With Clarithromycin and Ethambutol in Adult Patients With Treatment-refractory Mycobacterium Avium Complex-lung Disease (MAC-LD)
Brief Title: A Study of Bedaquiline Administered as Part of a Treatment Regimen With Clarithromycin and Ethambutol in Adult Patients With Treatment-refractory Mycobacterium Avium Complex-lung Disease (MAC-LD)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108897; TMC207NTM3002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2020-11-12; First posted 2020-11-16 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Treatment-refractory Mycobacterium Avium Complex-lung Disease (MAC-LD)
MeSH Terms: interventions — bedaquiline; Clarithromycin; Ethambutol; Rifampin; Rifabutin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A: Bedaquiline (BDQ) + Clarithromycin (CAM) + Ethambutol (EB) (Experimental): Participants will receive BDQ 400 milligrams (mg) (4*100 mg tablets) once daily (qd) from Week 1-2 (loading phase), BDQ 200 mg (2*100mg tablets) bi-weekly (biw) from Week 3 to 48 (maintenance phase) and CAM 400 mg or 500 mg twice daily (2*200 mg tablets) along with EB 500-750 mg or 15 mg/kg once a day or maximum daily dose of 1.0 gram for up to Week 48.
  Interventions: Drug: Bedaquiline; Drug: Clarithromycin; Drug: Ethambutol
- Group B: Rifampicin (RFP) or Rifabutin (RBT) + CAM + EB (Active Comparator): Participants will receive maximum of 4 capsules of RFP 450 mg daily (or maximum daily dose of 600 mg), CAM 400 mg or 500 mg (2*200 mg tablets) twice a day along with EB 500-750 mg daily or 15 mg/kg once a day or maximum daily dose of 1.0 gram for up to Week 48, followed by 2 capsules of RBT 300 mg or 150 mg once a day.
  Interventions: Drug: Clarithromycin; Drug: Ethambutol; Drug: Rifampicin; Drug: Rifabutin

INTERVENTIONS:
Drug: Bedaquiline — Participants will receive BDQ tablets only/
  Arms: Group A: Bedaquiline (BDQ) + Clarithromycin (CAM) + Ethambutol (EB)
Drug: Clarithromycin — Participants will receive CAM 400 or 500 mg twice a day.
Drug: Ethambutol — Participants will receive 500 to 750 mg daily (maximum daily dose of 1.0 gram [g]) or 15 mg/kg once a day.
Drug: Rifampicin — Participants will receive daily dose is 450 mg (maximum 600 mg) RFP capsule once a day.
  Arms: Group B: Rifampicin (RFP) or Rifabutin (RBT) + CAM + EB
Drug: Rifabutin — Participants will receive daily dose of RBT 300 mg or 150 mg capsules once a day.
  Arms: Group B: Rifampicin (RFP) or Rifabutin (RBT) + CAM + EB

SUMMARY:
The purpose of the study is to evaluate the efficacy of bedaquiline (BDQ) compared with rifamycin when administered as part of a treatment regimen with clarithromycin (CAM) and ethambutol (EB) in adult participants with treatment-refractory Mycobacterium avium complex-lung disease (MAC-LD) at Week 24 for microbiological assessment in mycobacteria growth indicator tube (MGIT).

ELIGIBILITY:
Inclusion Criteria:

* Has body weight greater than or equal to (>=) 40 kilograms (kg) at screening and on Day 1
* Has radiological evidence consistent with nontuberculous mycobacterial lung disease (NTM-LD) based on a chest Computed Tomography (CT) scan taken within 6 months prior to screening or at screening
* Has at least 2 positive sputum cultures of Mycobacterium avium complex (MAC) (sputum cultures to be taken at least 4 weeks apart): one obtained within 12 months prior to screening, which was documented while being treated for Mycobacterium avium complex lung disease (MAC-LD) for a total of at least 6 months; and one at screening (by central microbiology laboratory)
* Received at least 6 months of consecutive MAC-LD treatment (at least 2 antibiotics for MAC, including a macrolide), that is either ongoing or has stopped within 12 months prior to screening
* No presence of cognitive dysfunction that would impact the completion of the patient reported outcome (PRO) assessments

Exclusion Criteria:

* Had previous exposure to bedaquiline (BDQ)
* Has active Tuberculosis (TB) disease
* Has cystic fibrosis, medically unstable respiratory disease (for example, chronic obstructive pulmonary disease, bronchiectasis, asthma)
* Has one or more cavities >=2 centimeter (cm) in diameter on a chest CT scan taken within 6 months prior to screening or at screening
* Treatment already includes an injectable/inhaled aminoglycoside within 3 months prior to screening or the investigator deems the participant to be a candidate for an injectable/inhaled aminoglycoside during screening period or at Day 1

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2024-11-06 (Actual); Study Completion 2025-11-14 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Sputum Culture Conversion in Mycobacteria Growth Indicator Tube (MGIT) at Week 24 | Week 24
  Percentage of participant with sputum culture conversion (defined as 3 consecutive negative sputum cultures taken at least 25 days apart) in MGIT at Week 24 will be assessed.

SECONDARY OUTCOMES:
Percentage of Participants with Sputum Culture Conversion in 7H10 or 7H11 agar media at Week 24 | Up to Week 24
  Percentage of participants with sputum culture conversion (defined as 3 consecutive negative sputum cultures taken at least 25 days apart) in 7H10 or 7H11 agar media at Week 24 will be assessed.
Change from Baseline in Patient-reported Health Status on Total Score of St. George's Respiratory Questionnaire (SGRQ) at Week 24 | Baseline and Week 24
  The SGRQ is a self-administered questionnaire that has been validated in participants with airways disease, specifically in participants with bronchiectasis. The SGRQ assesses health-related quality of life in participants with chronic pulmonary disease by evaluating 3 health domains: symptoms (distress caused by respiratory symptoms); activity (effects of disturbances on mobility and physical activity); and impacts (the effect of disease on factors such as employment, personal control of one's health, and need for medication). A composite total score is derived as the sum of domain scores for symptoms, activity, and impact (0 = best possible score and 100 = worst possible score).
Percentage of Participants with Sputum Culture Conversion in MGIT and 7H10 or 7H11 agar media at Week 48 and Week 60 | Up to Week 48 and Week 60
  Percentage of participants with sputum culture conversion (defined as 3 consecutive negative sputum cultures taken at least 25 days apart) in MGIT and 7H10 or 7H11 agar media at Week 48 and Week 60 will be assessed.
Percentage of Participants with Sputum Culture Negativity in MGIT and 7H10 or 7H11 at each visit after Week 2 | From Week 2 to Week 60
  Percentage of participants with sputum culture negativity in MGIT and 7H10 or 7H11 at each visit after Week 2 will be assessed.
Time to Sputum Culture Conversion in MGIT up to Week 48 | Up to Week 48
  Sputum culture conversion is defined as 3 consecutive negative sputum cultures taken at least 25 days apart. Percentage of participants with sputum culture in 7H10 or 7H11 agar media at Week 24 will be assessed. Time to sputum culture conversion in MGIT up to Week 48 will be assessed.
Time to Positivity in MGIT up to Week 48 | Up to Week 48
  Time to positivity in MGIT up to week 48 will be assessed.
Change From Baseline in Patient Reported Health Status on Total Score of SGRQ at Weeks 48 and 60 | From baseline to Week 48 and Week 60
  The SGRQ is a self-administered questionnaire that has been validated in participants with airways disease, specifically in participants with bronchiectasis. The SGRQ assesses health-related quality of life in participants with chronic pulmonary disease by evaluating 3 health domains: symptoms (distress caused by respiratory symptoms); activity (effects of disturbances on mobility and physical activity); and impacts (the effect of disease on factors such as employment, personal control of one's health, and need for medication). A composite total score is derived as the sum of domain scores for symptoms, activity, and impact (0 = best possible score and 100 = worst possible score). A within patient reduction from baseline in score of 4 units is generally recognized as a clinically meaningful improvement in quality of life.
Change From Baseline in Lung Function Parameters (Forced Vital Capacity) at Weeks 24, 48, and 60 | At Weeks 24, 48, and 60
  The lung function parameters including forced expiration volume will be assessed.
Change From Baseline in Lung Function Parameters (Inspiratory Capacity) at Weeks 24, 48, and 60 | At Weeks 24, 48, and 60
  The lung function parameters including Inspiratory Capacity will be assessed.
Change From Baseline in Lung Function Parameters (Functional Residual Capacity and Total Lung Capacity) at Weeks 24, 48, and 60 | At Weeks 24, 48, and 60
  The lung function parameters including functional residual capacity and total lung capacity will be assessed.
Percentage of Participants who Undergo a Change in Their Mycobacterium Avium Complex-lung Disease (MAC-LD) Treatment Regimen by Week 24 and by Week 48 in Group A and by Week 60 in Group B | Week 24 and Week 48 (Group A) and by week 60 (Group B)
  Percentage of participants who undergo a change in their MAC-LD treatment regimen will be assessed.
Number of Participants with Adverse Events (AE) | Up to Week 60
  An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non-investigational) product, whether or not related to that medicinal (investigational or non-investigational) product.
Number of Participants with Clinical Laboratory Abnormalities | Up to Week 60
  Number of participants with clinical laboratory abnormalities (Hematology, Clinical chemistry, and Urinalysis) will be assessed.
Number of Participants with 12-Lead Electrocardiogram (ECG) Abnormalities | Up to Week 60
  Number of participants with 12-Lead ECG Abnormalities will be assessed.
Number of Participants with Vital Signs Abnormalities | Up to Week 60
  Number of participants with vital signs abnormalities (body temperature [axillary], heart rate, respiratory rate, oxygen saturation, blood pressure [systolic and diastolic]) will be assessed.
Number of Participants with Physical Examination Abnormalities | Up to Week 60
  Number of Participants with physical examination abnormalities (all body systems [including height and body weight measurement] and observation for skin events/reactions) will be assessed.
Number of Participants with Visual Examination Abnormalities | Up to Week 60
  Number of participants with visual examination abnormalities (visual acuity testing, color discrimination, visual field testing, and fundoscopy and audiology) will be assessed.
Maximum Plasma Concentration (Cmax) of Bedaquiline and its Metabolite M2 | Day 1, Weeks 2, 8, 12, 24 and Week 48
  Cmax is defined as maximum observed analyte concentration.
Minimum Plasma Concentration Between 0 Hour and the Dosing Interval (tau) (Ctrough) of Bedaquiline and its Metabolite M2 | Day 1, Weeks 2, 8, 12, 24 and Week 48
  Ctrough is the minimum plasma concentration between 0 hour and dosing interval (tau).
Area Under the Plasma Concentration-time Curve From Time Zero to End of Dosing Interval (tau) (AUC [0-tau]) of Bedaquiline and its Metabolite M2 | Day 1, Weeks 2, 8, 12, 24 and Week 48
  AUC (0-tau) is area under the plasma concentration-time curve from time zero to end of dosing interval (tau).
Cmax of Clarithromycin and its Metabolite 4-OH CAM | Day 1, Weeks 2, 8, 12 and 24
  Cmax is defined as maximum observed analyte concentration.
C (0-trough) of Clarithromycin and its Metabolite 4-OH CAM | Day 1, Weeks 2, 8, 12 and 24
  Ctrough is the minimum plasma concentration between 0 hour and dosing interval (tau).
AUC (0-tau) of Clarithromycin and its Metabolite 4-OH CAM | Day 1, Weeks 2, 8, 12 and 24
  AUC (0-tau) is area under the plasma concentration-time curve from time zero to end of dosing interval (tau).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan clinical Trials, Study Director — Janssen Pharmaceutical K.K.
Locations (55):
- Japan (47):
  - Fukuoka University Chikushi Hospital, Chikushino-shi
  - St. Luke's International Hospital, Chūōku
  - Fukui Prefectural Hospital, Fukui-shi
  - National Hospital Organization Ibarakihigashi, Funaishikawa
  - Gifu Prefectural General Medical Center, Gifu
  - Hamamatsu Rosai Hospital, Hamamatsu
  - Seirei Hamamatsu General Hospital, Hamamatsu
  - National Hospital Organization Tenryu Hospital, Hamamatue
  - Matsunami General Hospital, Hashima-gun
  - Matsunami Health Promotion Clinic, Hashimagun Kasamatsucho
  - National Hospital Organization Himeji Medical Center, Himeji
  - Saitama Medical University Hospital, Iruma-gun
  - National Hospital Organization Minami Kyoto Hospital, Jōyō
  - Fukujuji Hospital, Kiyose
  - Kobe City Medical Center West Hospital, Kobe Nagata-Ku
  - National Hospital Organization Kochi National Hospital, Kochi
  - National Hospital Organization Fukuoka Higashi Medical Center, Koga
  - Saitama Prefectural Cardiovascular and Respiratory Center, Kumagaya
  - Rakuwakai Otowa Hospital, Kyoto
  - National Hospital Organization Kyoto Medical Center, Kyoto
  - Matsusaka Municipal Hospital, Matsusaka
  - Musashino Red Cross Hospital, Musashino
  - Nagaoka Red Cross Hospital, Nagaoka
  - Nagasaki University Hospital, Nagasaki
  - Kojunkai Daido Clinic, Nagoya
  - National Hospital Organization Nagoya Medical Center, Nagoya
  - National Hospital Organization Nishiniigata Chuo Hospital, Niigata
  - National Hospital Organization Omuta Hospital, Omuta
  - National Hospital Organization Sagamihara National Hospital, Sagamihara
  - Saitama City Hospital, Saitama-shi
  - Kinki-chuo Chest Medical Center, Sakai
  - Hokkaido Medical Center, Sapporo Nishi-Ku
  - Tohoku Medical And Pharmaceutical University Hospital, Sendai
  - National Hospital Organization Nara Medical Center, Shichijō
  - Tokyo Shinagawa Hospital, Shinagawa-ku
  - National Center for Global Health and Medicine, Shinjuku
  - Keio University Hospital, Shinjuku-ku
  - Nagano Prefectural Shinshu Medical Center, Suzaka
  - National Hospital Organization Tokyo Medical Center, Tokyo
  - National Hospital Organization Tokyo National Hospital, Tokyo
  - National Hospital Organization Osaka Toneyama Medical Center, Toyonaka-shi
  - Toyota Kosei Hospital, Toyota
  - Toyota Memorial Hospital, Toyota-shi
  - National Hospital Organization Ehime Medical Center, Tōon
  - JRC Wakayama Medical Center, Wakayama
  - Shimonoseki City Hospital, Yamaguchi
  - Kanagawa Cardiovascular And Respiratory Center, Yokohama
- South Korea (4):
  - Chonnam National University Hospital, Gwangju
  - The Catholic University of Korea, Incheon St. Mary's Hospital, Incheon
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Taiwan (4):
  - Kaohsiung Medical University Chung Ho Memorial Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency